CLINICAL TRIAL: NCT00116194
Title: Physical Exercise to Prevent Disability Pilot Study
Brief Title: The LIFE Study: Lifestyle Interventions and Independence for Elders, Pilot
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AG0021; U01AG022376 (NIH)
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2008-12

CONDITIONS: Physically Challenged; Aging
Keywords: exercise; activities of daily living; ADL; loss of mobility; risk of disability; physical activity; mobility disability
MeSH Terms: conditions — Motor Activity | interventions — Exercise

INTERVENTIONS:
Behavioral: Physical Activity

SUMMARY:
The purpose of this study is to gather preliminary data that will determine the feasibility of conducting a Phase III, randomized, controlled trial (RCT) that will provide definite evidence in the use of physical exercise to prevent mobility disability in older persons.

DETAILED DESCRIPTION:
As the life expectancy of older Americans increases, prevention of age-associated physical function decline and disabilities has emerged as a major clinical and public health priority. A critical factor in an older person's ability to function independently is mobility, the ability to move without assistance. Older people who lose mobility are less likely to remain in the community, have higher rates of morbidity, mortality, and hospitalizations and experience a poorer quality of life. While several studies suggest that physical activity may prevent physical disability, including mobility disability in both healthy and frail older adults, definitive evidence is lacking. A Phase 3, randomized, controlled trial is needed to fill this evidence gap. Currently data to estimate sample size needs for such a trial are insufficient and further feasibility data should be gathered before such a trial can be effectively designed and implemented.

To refine key trial design benchmarks (including sample size calculations to demonstrate the feasibility of a full-scale trial and refining/developing recruitment, procedures, materials and organizational infrastructure), the LIFE (Lifestyle Interventions for Independence in Elders) study conducts a pilot, single-blind, randomized, controlled trial involving comparison of a physical activity program of moderate intensity to a successful aging program. Approximately 400 sedentary persons aged 70 to <90 years who are at risk of disability are followed for at least one year at four intervention sites: Wake Forest University School of Medicine in Winston Salem, NC; the University of Pittsburgh in Pittsburgh, PA; the Cooper Institute in Dallas, TX; and the Stanford University in Palo Alto, CA. The Administrative Coordinating Center and the Data Management and Quality Control Center are at Wake Forest University School of Medicine.

The LIFE study assesses the combined outcome of major mobility disability, defined as the incapacity to walk 400 meters (m), or death, which will be the primary outcome of the full-scale study. This outcome has not been used in previous randomized, controlled trials, and therefore, a pilot study is needed to assess its incidence rate. Secondary outcomes include ADL disability, major fall injuries and cardiovascular events. LIFE explores the effects of the intervention on physical performance measures, cognitive function, health-related quality of life, and use of health care services. In addition, LIFE explores and performs cost-effectiveness analyses of the intervention.

This pilot study will yield the necessary preliminary data to design a definitive Phase 3, randomized, controlled trial. By providing a conclusive answer regarding whether physical activity is effective for preventing major mobility disability or death, the results of the full-scale trial will have relevant clinical and public health implications, and will fill an important gap in knowledge for practicing evidence-based geriatric medicine.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 70 to 89
* Residency in the area for at least 9 months in the next year
* Summary score of under 10 on the Established Populations for Epidemiologic Studies of the Elderly (EPESE) physical performance battery; ability to complete the 400 m walk test within 15 minutes without sitting and without the use of an assistive device (including a cane) or the help of another person
* Able to understand and perform the required study procedures; no diagnosis of dementia
* Sedentary lifestyle, i.e., has spent less than 20 minutes per week in the past month getting regular physical activity
* Willing to give informed consent, willing to be randomized to either intervention, and to follow the protocol for the group to which they have been assigned
* Successful completion of the behavioral run-in

Exclusion Criteria:

* Potential difficulty adhering to either intervention
* Unable or unwilling to give informed consent or accept randomization
* Participation may be unsafe
* Serious health conditions that would interfere with the intervention goals
* Already physically active to a degree that the adoption of an activity program would be of little additional benefit
* Self-reported inability to walk two blocks
* Use of walker or assistive device to complete the 400 m walk

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 424
Dates: Start 2004-04; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Combined outcome of ability to walk 400 m without the use of an assistive device or adjudicated evidence of inability to walk 400 m or death
Drop-in, drop-out, and loss to follow-up rates
Established Populations for Epidemiologic Studies of the Elderly (EPESE) physical performance score
4 m gait speed
400 m gait speed
Self-reported disability scale

SECONDARY OUTCOMES:
Onset of self- or proxy-reported and objectively assessed disability in activities of daily living (ADLs)
Serious fall injuries
Combined cardiovascular events
Acute care hospitalizations and nursing home admissions
Cognitive function measures; Health-related quality of life (HRQL), as reflected by depressive symptoms, anxiety, energy and fatigue level, sleep, and pain; Nursing home and acute-care hospitalization length of stay; Cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pahor, MD, Principal Investigator — Professor and Chair, Department of Aging and Geriatric Research, College of Medicine, Director Institute on Aging, University of Florida; Jack Guralnik, MD, PhD, Principal Investigator — Acting Chief, Laboratory of Epidemiology, Demography and Biometry, National Institute on Aging
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Cooper Institute, Dallas, Texas

REFERENCES:
- [Background] Rejeski WJ, Fielding RA, Blair SN, Guralnik JM, Gill TM, Hadley EC, King AC, Kritchevsky SB, Miller ME, Newman AB, Pahor M. The lifestyle interventions and independence for elders (LIFE) pilot study: design and methods. Contemp Clin Trials. 2005 Apr;26(2):141-54. doi: 10.1016/j.cct.2004.12.005. PMID 15837437
- [Background] Guralnik JM, LaCroix AZ, Abbott RD, Berkman LF, Satterfield S, Evans DA, Wallace RB. Maintaining mobility in late life. I. Demographic characteristics and chronic conditions. Am J Epidemiol. 1993 Apr 15;137(8):845-57. doi: 10.1093/oxfordjournals.aje.a116746. PMID 8484376
- [Background] Tinetti ME, Baker DI, McAvay G, Claus EB, Garrett P, Gottschalk M, Koch ML, Trainor K, Horwitz RI. A multifactorial intervention to reduce the risk of falling among elderly people living in the community. N Engl J Med. 1994 Sep 29;331(13):821-7. doi: 10.1056/NEJM199409293311301. PMID 8078528
- [Background] Ettinger WH Jr, Burns R, Messier SP, Applegate W, Rejeski WJ, Morgan T, Shumaker S, Berry MJ, O'Toole M, Monu J, Craven T. A randomized trial comparing aerobic exercise and resistance exercise with a health education program in older adults with knee osteoarthritis. The Fitness Arthritis and Seniors Trial (FAST). JAMA. 1997 Jan 1;277(1):25-31. PMID 8980206
- [Background] Penninx BW, Messier SP, Rejeski WJ, Williamson JD, DiBari M, Cavazzini C, Applegate WB, Pahor M. Physical exercise and the prevention of disability in activities of daily living in older persons with osteoarthritis. Arch Intern Med. 2001 Oct 22;161(19):2309-16. doi: 10.1001/archinte.161.19.2309. PMID 11606146
- [Result] LIFE Study Investigators; Pahor M, Blair SN, Espeland M, Fielding R, Gill TM, Guralnik JM, Hadley EC, King AC, Kritchevsky SB, Maraldi C, Miller ME, Newman AB, Rejeski WJ, Romashkan S, Studenski S. Effects of a physical activity intervention on measures of physical performance: Results of the lifestyle interventions and independence for Elders Pilot (LIFE-P) study. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1157-65. doi: 10.1093/gerona/61.11.1157. PMID 17167156
- [Derived] Ip EH, Chen SH, Rejeski WJ, Bandeen-Roche K, Hayden KM, Hugenschmidt CE, Pierce J, Miller ME, Speiser JL, Kritchevsky SB, Houston DK, Newton RL, Rapp SR, Kitzman DW. Gradient and Acceleration of Decline in Physical and Cognitive Functions in Older Adults: A Disparity Analysis. J Gerontol A Biol Sci Med Sci. 2022 Aug 12;77(8):1603-1611. doi: 10.1093/gerona/glac109. PMID 35562076
- [Derived] Fielding RA, Guralnik JM, King AC, Pahor M, McDermott MM, Tudor-Locke C, Manini TM, Glynn NW, Marsh AP, Axtell RS, Hsu FC, Rejeski WJ; LIFE study group. Dose of physical activity, physical functioning and disability risk in mobility-limited older adults: Results from the LIFE study randomized trial. PLoS One. 2017 Aug 18;12(8):e0182155. doi: 10.1371/journal.pone.0182155. eCollection 2017. PMID 28820909
- [Derived] Newman AB, Dodson JA, Church TS, Buford TW, Fielding RA, Kritchevsky S, Beavers D, Pahor M, Stafford RS, Szady AD, Ambrosius WT, McDermott MM; LIFE Study Group. Cardiovascular Events in a Physical Activity Intervention Compared With a Successful Aging Intervention: The LIFE Study Randomized Trial. JAMA Cardiol. 2016 Aug 1;1(5):568-74. doi: 10.1001/jamacardio.2016.1324. PMID 27439082
- [Derived] Dotson VM, Hsu FC, Langaee TY, McDonough CW, King AC, Cohen RA, Newman AB, Kritchevsky SB, Myers V, Manini TM, Pahor M; LIFE STUDY GROUP. Genetic Moderators of the Impact of Physical Activity on Depressive Symptoms. J Frailty Aging. 2016;5(1):6-14. doi: 10.14283/jfa.2016.76. PMID 26980363
- [Derived] O'Hartaigh B, Pahor M, Buford TW, Dodson JA, Forman DE, Gill TM; LIFE Study Group. Physical activity and resting pulse rate in older adults: findings from a randomized controlled trial. Am Heart J. 2014 Oct;168(4):597-604. doi: 10.1016/j.ahj.2014.07.024. Epub 2014 Jul 30. PMID 25262271
- [Derived] Heffernan KS, Manini TM, Hsu FC, Blair SN, Nicklas BJ, Kritchevsky SB, Newman AB, Sutton-Tyrrell K, Church TS, Haskell WL, Fielding RA. Relation of pulse pressure to long-distance gait speed in community-dwelling older adults: findings from the LIFE-P study. PLoS One. 2012;7(11):e49544. doi: 10.1371/journal.pone.0049544. Epub 2012 Nov 21. PMID 23185357
- [Derived] Houston DK, Tooze JA, Hausman DB, Johnson MA, Nicklas BJ, Miller ME, Neiberg RH, Marsh AP, Newman AB, Blair SN, Kritchevsky SB. Change in 25-hydroxyvitamin D and physical performance in older adults. J Gerontol A Biol Sci Med Sci. 2011 Apr;66(4):430-6. doi: 10.1093/gerona/glq235. Epub 2011 Feb 16. PMID 21325343
- [Derived] Hsu FC, Rejeski WJ, Ip EH, Katula JA, Fielding R, Jette AM, Studenski SA, Blair SN, Miller ME. Evaluation of the late life disability instrument in the Lifestyle Interventions and Independence for Elders Pilot (LIFE-P) study. Health Qual Life Outcomes. 2010 Oct 6;8:115. doi: 10.1186/1477-7525-8-115. PMID 20925931
- See also: The LIFE Study — https://www.thelifestudy.org/public/index.cfm